CLINICAL TRIAL: NCT06027177
Title: P4D - Personalized, Predictive, Precise & Preventive Medicine for Major Depression
Brief Title: Personalized, Predictive, Precise & Preventive Medicine for Major Depression
Acronym: P4D
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: University Medicine Greifswald (Other); Wuerzburg University Hospital (Other); Goethe University (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Other Study IDs: P4D_cohort; DRKS00032215 (Registry Identifier: DRKS German Clinical Trials Register)
Record Dates: First submitted 2023-08-22; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder; Persistent Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are used for a variety of purposes. In addition to standard clinical laboratory tests, genetic (nanopore sequencing) and epigenetic (miRNA, methylation) tests will be performed. In addition, drug levels will be monitored regularly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depressive disorders are among the most common psychiatric disorders. However, this disorder is multifaceted, as are its etiological factors, and is not yet fully understood. Within the framework of the P4D study, 1000 patients with depression will be comprehensively examined. In addition to the recording of psychological factors by means of questionnaires and third-party assessments, imaging and electrophysiological procedures (functional and structural MRI, EEG) are used to assess brain structure and function. In addition, blood is drawn from the subjects to analyze these samples for various biological markers (e.g., genetics). Drug level measurements are also performed.

The goal is to perform an in-depth characterization (phenotyping) of individuals with a depressive disorder. These findings could be used to individualize and improve therapy for depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* MDD: ICD-10: F32.1-3, F33.1-3 first or recurrent depressive episode (confirmed by MINI-DIPS) and/or PDD: F34.1
* Symptom severity: Moderate to severe (MADRS ≥ 20).
* First depressive episode before 50 years of age
* Signed informed consent form
* Capacity to consent

Exclusion Criteria:

* Acute Suicidality
* Placement according to state law (e.g. §16/17 Nds. PsychKG)
* The following diagnoses in the life course: Dementia, schizophrenia, schizoaffective disorder, bipolar disorder, substance dependence with currently necessary detoxification
* Concurrent participation in other clinical trials that are not being conducted within the framework of the P4D project

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe depressive disorder, aged between 18 and 70 years, who are undergoing inpatient treatment will be recruited. Patients should fulfil the inclusion criteria. All patients who meet the criteria are given information by a doctor and have the opportunity to ask further questions. Their participation in the study is voluntary and they give their written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Remission after 7 weeks of treatment | Baseline and Follow-up (Week 7)
  The Montgomery-Asberg-Depression-Scale (MADRS) is used to measure the severity of depressive symptoms. A score lower 7 is the cut-off.

SECONDARY OUTCOMES:
Recording of psychometric changes in the clinical course of treatment | Baseline and Follow-up (Week 7)
  A range of psychometric information is collected. These include questionnaires, third party ratings and a cognitive assessment, as well as neuroimaging (functional and structural MRI), neurophysiology (EEG) and polysomnography (PSG).
Frequency of other concomitant treatments (e.g., additional psychotherapeutic treatment) | Follow-up (Week 7)
  Psychotherapy sessions (individual and group therapy) are recorded for 7 weeks. Alternative treatments (e.g. transcranial magnetic stimulation and electroconvulsive therapy) are also recorded.
Treatment/study dropout rates | Drop-out rates are collected throughout the data collection period, over two years. Starting at study enrollment of the first subject until complete completion of the last subject.
  Dropout rates are recorded with reasons.
Attitudes (acceptance, fears, and prejudices) regarding biomarker-guided examinations and technical procedures among the population | The survey will be conducted over a 2-week period in late August / early September 2023.
  Representative population survey
Patient-doctor relationship | Baseline and Follow-up (Week 7)
  The Patient-Doctor-Relationship-Questionnaire (PDRQ-9) is used to assess the quality of the therapeutic relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Helge Frieling, Prof. Dr.med, Study Chair — Hannover Medical School

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is planned.
Time Frame: Data will be kept pseudonymised for 10 years and then anonymised.
Access Criteria: Upon individual request, data may be made available before this time.